CLINICAL TRIAL: NCT03088878
Title: A Phase 1b/2 Study of the ROR1-Targeting Monoclonal Antibody, Cirmtuzumab (UC-961), and the Bruton Tyrosine Kinase Inhibitor, Ibrutinib, in Patients With B-Cell Lymphoid Malignancies
Brief Title: A Study of Cirmtuzumab and Ibrutinib in Patients With B-Cell Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncternal Therapeutics, Inc (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); University of California, San Diego (Other); Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIRM-0001 (CIRLL); NCT03420183 (obsolete NCT alias)
Record Dates: First submitted 2017-03-02; First posted 2017-03-23 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma
Keywords: Chronic lymphocytic leukemia; Small lymphocytic lymphoma; Mantle cell lymphoma; Receptor Tyrosine Kinase-like Orphan Receptor 1 (ROR1); Bruton Tyrosine Kinase (BTK); Ibrutinib; Marginal zone lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — cirmtuzumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Cirmtuzumab followed by Cirmtuzumab plus ibrutinib
  Interventions: Drug: Cirmtuzumab (2-16 kg/mg) plus Ibrutinib; Drug: Cirmtuzumab (300mg) plus Ibrutinib; Drug: Cirmtuzumab (600 mg) plus ibrutinib
- Part 2 (Experimental): Cirmtuzumab plus ibrutinib
  Interventions: Drug: Cirmtuzumab (RDR) plus ibrutinib
- Part 3 - Arm A (Experimental): Cirmtuzumab plus ibrutinib
  Interventions: Drug: Cirmtuzumab plus ibrutinib
- Part 3 - Arm B (Active Comparator): Ibrutinib only
  Interventions: Drug: Ibrutinib alone

INTERVENTIONS:
Drug: Cirmtuzumab (2-16 kg/mg) plus Ibrutinib — Participants will receive escalating doses of cirmtuzumab (2-16 mg/kg) administered IV every 2 weeks for 5 administrations and then every 4 weeks thereafter, plus ibrutinib (420 or 560 mg) orally once daily, starting at week 4.
  Other Names: UC-961; Imbruvica
  Arms: Part 1
Drug: Cirmtuzumab (300mg) plus Ibrutinib — Participants will receive cirmtuzumab (300 mg) administered IV every 2 weeks for 5 administrations and then every 4 weeks thereafter, plus ibrutinib (420 mg) orally once daily.
  Other Names: UC-961; Imbruvica
  Arms: Part 1
Drug: Cirmtuzumab (600 mg) plus ibrutinib — Participants will receive cirmtuzumab (600 mg) administered IV every 2 weeks for 5 administrations and then every 4 weeks thereafter, plus ibrutinib (420 mg) orally once daily.
  Other Names: UC-961; Imbruvica
  Arms: Part 1
Drug: Cirmtuzumab (RDR) plus ibrutinib — Participants will receive cirmtuzumab (600 mg) administered IV every 2 weeks for 3 administrations and then every 4 weeks thereafter, plus ibrutinib (420 or 560 mg) orally once daily
  Other Names: UC-961; Imbruvica
  Arms: Part 2
Drug: Cirmtuzumab plus ibrutinib — Arm A: Participants will receive cirmtuzumab (600 mg) administered IV every 2 weeks for 3 administrations and then every 4 weeks thereafter, plus ibrutinib (420 mg) orally once daily.
  Other Names: UC-961; Imbruvica
  Arms: Part 3 - Arm A
Drug: Ibrutinib alone — Arm B: Participants will receive ibrutinib (420 mg) orally once daily
  Other Names: Imbruvica
  Arms: Part 3 - Arm B

SUMMARY:
This is Phase 1b/2 study to investigate the safety and effectiveness of the investigational drug, cirmtuzumab, when given in combination with ibrutinib in patients with B-cell lymphoid malignancies. Cirmtuzumab is a monoclonal antibody that attaches to a protein (called ROR 1) that is found on hematologic tumor cells. ROR1 has been shown to play a role in cell signaling that cause leukemia and lymphoma cells to grow and survive. ROR1 is rarely found on healthy cells.

DETAILED DESCRIPTION:
This is a Phase 1b/2 study to investigate the safety and effectiveness of the investigational drug, cirmtuzumab (INN:zilovertamab), when given in combination with ibrutinib in patients with B-cell lymphoid malignancies. The Phase 1b will be conducted in two parts (Part 1 and Part 2). Part 1 is a dose-finding evaluation of the sequential administration of cirmtuzumab monotherapy followed by cirmtuzumab and ibrutinib combination therapy in chronic lymphocytic leukemia /small lymphocytic leukemia (CLL/SLL), previously treated mantle cell lymphoma (MCL) subjects that are BTKI naiive or have received a prior Bruton tyrosine kinase (BTK) inhibitor therapy, unless they demonstrated primary or acquired resistance to BTKi. Up to 48 subjects will be enrolled in Part 1 to determine the recommended dosing regimen (RDR). In Part 2, up to 60 subjects (CLL/SLL, MCL and MZL (marginal zone lymphoma) will be enrolled to further evaluate the safety and pharmacology of the cirmtuzumab and ibrutinib combination given at the RDR determined in Part 1 of the study. MZL subjects that have been previously treated and have relapsed after or progressed during at least one prior anti-CD20 -based therapy will be evaluated. In the Phase 2 (Part 3) portion of the study, approximately 30 subjects with CLL/SLL who may have received minimal prior BTK inhibitor therapy will be randomized to either Arm 1 (cirmtuzumab and ibrutinib) at the RDR or Arm 2 (ibrutinib alone) to evaluate the clinical activity and safety of the two arms.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of age ≥18 years.
2. ECOG performance status of 0, 1, or 2
3. Histological diagnosis of CLL/SLL, MCL or MZL (including splenic,nodal and extranodal subtypes) as documented in medical records (pathology reports and slides or blocks should be available for review or additional testing).
4. MCL has been previously treated and has relapsed after or progressed during prior therapy. CLL/SLL may have been previously treated or are treatment naïve but now require therapy. MZL has been previously treated and has relapsed after or progressed during at least one prior anti-CD20 -based therapy
5. A medically appropriate candidate for ibrutinib treatment (based on the judgement of the clinical investigator).
6. Patients who have received prior BTK inhibitor therapy are eligible, unless they demonstrated primary or acquired resistance to a BTK inhibitor or experienced a serious or severe adverse event attributed to BTK inhibitor therapy.
7. Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥1 non-biopsied, non-irradiated lesion that measures >1.5 cm in the longest dimension [LD] and ≥1.0 cm in the longest perpendicular dimension [LPD] as assessed by computed tomography [CT] or magnetic resonance imaging [MRI]).
8. Current medical need for therapy due to disease-related symptoms, lymphadenopathy, organomegaly, extranodal organ involvement, or progressive disease.
9. Completion of all previous therapy (including any Bcl-2 or PI3K inhibitor therapy, surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥1 week (or ≥3 half-lives of the previous drug) before the start of study therapy.
10. All acute toxic effects of any prior antitumor therapy resolved to Grade ≤1 before the start of study therapy (with the exceptions of alopecia, or neurotoxicity [Grade 1 or 2 permitted], or selected laboratory parameters [Grade 1 or Grade 2 permitted with exceptions as noted below]).
11. Adequate bone marrow function:

    1. Absolute neutrophil count (ANC) ≥1.0 × 109/L.
    2. Platelet count ≥50 × 109/L.
    3. Hemoglobin ≥8.0 g/dL maintained for ≥1 week from any prior transfusion.
12. Adequate hepatic profile:

    1. Serum alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN).
    2. Serum aspartate aminotransferase (AST) ≤3 × ULN.
    3. Serum bilirubin ≤1.5 × ULN unless elevated due to Gilbert syndrome.
13. Adequate renal function:

    1. Estimated creatinine clearance (eClCR) >30 mL/minute (with eClCR to be calculated by the Cockcroft-Gault formula [see Appendix 12.2]), or
    2. Measured creatinine clearance >30 mL/minute (as assessed with a 24-hour urine collection).
14. Adequate coagulation profile:

    1. Prothrombin time (PT) ≤1.5 × ULN.
    2. Activated partial thromboplastin time (aPTT) ≤1.5 × ULN.
15. Negative viral serology:

    1. Negative human immunodeficiency virus (HIV) antibody.
    2. Negative hepatitis B surface antigen (HBsAg) and negative hepatitis B core (HBc) antibody or undetectable hepatitis B (HBV) deoxyribonucleic acid (DNA) by quantitative polymerase chain reaction (PCR) testing.
    3. Negative hepatitis C virus (HCV) antibody or negative HCV RNA by quantitative PCR.
16. For female patients of childbearing potential, a negative urine or serum pregnancy test prior to the start of study therapy.
17. For female patients of childbearing potential, willingness to use a highly effective method of contraception from the start of the screening period until ≥3 months after the last dose of cirmtuzumab and ≥1 month after the last dose of ibrutinib, whichever is later. Note: A female patient is considered to be of childbearing potential unless she has had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy; has medically documented ovarian failure (with serum estradiol and follicle-stimulating hormone [FSH] levels within the institutional laboratory postmenopausal range and a negative serum or urine beta human chorionic gonadotropin [βHCG]); or is menopausal (age ≥50 years with amenorrhea for ≥6 months).
18. For male patients who can father a child and are having intercourse with females of childbearing potential who are not using adequate contraception, willingness to use an effective method of contraception from the start of study therapy until ≥3 months after the last dose of cirmtuzumab and ≥3 months after the last dose of ibrutinib, whichever is later and to refrain from sperm donation from the start of study therapy until ≥3 months after administration of the final dose of either of the study drugs. Note: A male patient is considered able to father a child unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy.
19. In the judgment of the investigator, participation in the protocol offers an acceptable benefit-to-risk ratio when considering current disease status, medical condition, and the potential benefits and risks of alternative treatments for the patient's cancer.
20. Willingness and ability of the patient to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions.
21. Evidence of a personally signed informed consent indicating that the patient is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

1. Known histological transformation to an aggressive lymphoma (ie, Richter transformation).
2. Known central nervous system malignancy.
3. Presence of another cancer with disease manifestations or therapy that could adversely affect subject safety or longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
4. Significant cardiovascular disease (eg, myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to start of study therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; or uncontrolled Grade ≥3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg) despite antihypertensive therapy.
5. Significant screening ECG abnormalities, including unstable cardiac arrhythmia requiring medication, atrial fibrillation/flutter, left bundle branch block, 2nd-degree atrioventricular (AV) block type II, 3rd-degree AV block, or Grade ≥2 bradycardia.
6. Gastrointestinal disease (eg, gastric or intestinal bypass surgery, pancreatic enzyme insufficiency, malabsorption syndrome, symptomatic inflammatory bowel disease, chronic diarrheal illness, bowel obstruction) that might interfere with drug absorption or with interpretation of gastrointestinal AEs.
7. Contraindication for ibrutinib use because of bleeding diathesis.
8. Evidence of an ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections) at the time of start of study therapy. Note: Patients with localized fungal infections of skin or nails are not precluded from participation.
9. In patients with prior hematopoietic progenitor cell transplantation, evidence of ongoing graft-versus-host disease (GVHD).
10. Pregnancy or breastfeeding.
11. Major surgery within 4 weeks before the start of study therapy.
12. Prior solid organ transplantation.
13. Prior anti-ROR1 therapy within 12 weeks prior to the start of study therapy.
14. Use of a moderate or strong inhibitor or inducer of cytochrome P450 (CYP) 3A4 within 7 days prior to the expected start of ibrutinib therapy.
15. Concurrent participation in another therapeutic or imaging clinical trial.
16. Any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a subject's ability to provide informed consent, adversely affect the subject's ability to cooperate and participate in the study, or compromise the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Choi, MD, Principal Investigator — University of California, San Diego
Locations (12):
- United States (12):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Sanford Stem Cell Clinical Center at UCSD, La Jolla, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Yale Cancer Center, New Haven, Connecticut
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Louisiana State University Health New Orleans (NCI Community Oncology Research Program), New Orleans, Louisiana
  - Hackensack Meridian Health, John Theurer Cancer Center, Hackensack, New Jersey
  - Northwell Health, New Hyde Park, New York
  - Manhattan Hematology Oncology Research Foundation, Inc., New York, New York
  - Columbia University Medical Center, New York, New York
  - The Christ Hospital Lindner Research Center, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557

RESULTS

PARTICIPANT FLOW:
Groups:
- MCL Phase 1b, Part 1: 2mg/kg; MCL Phase 1b, Part 1: 4mg/kg; MCL Phase 1b, Part 1: 8mg/kg; MCL Phase 1b, Part 1: 16 mg/kg; MCL Phase 1b, Part 2: 600 mg; CLL Phase 1b, Part 1: 2 mg/kg; CLL Phase 1b, Part 1: 4 mg/kg; CLL Phase 1b, Part 1: 8 mg/kg; CLL Phase 1b, Part 1: 16 mg/kg; CLL Phase 1b, Part 1: 300 mg; CLL Phase 1b, Part 1: 600 mg; CLL Phase 1b, Part 2: 600mg: Part 1:
  * Cirmtuzumab given by IV infusion every 2 weeks for 5 administrations (Weeks 0, 2, 4, 6, 8) and then every 4 weeks thereafter (Weeks 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52) at a dose of either 2, 4, 8, or 16 mg/kg. After establishment of safety at these dose levels, fixed doses of 300 and 600 mg IV per dose will be examined in patients with CLL/SLL.
  * Ibrutinib self-administered orally, QD, continuously starting in Week 4 at a dose of either 420 mg/day (for patients with CLL/SLL) or at a dose of 560 mg/day (for patients with MCL).
  Part 2:
  * Cirmtuzumab given by IV infusion every 2 weeks for 3 administrations (Weeks 0, 2, 4) and then every 4 weeks thereafter (Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52) using the RDR of cirmtuzumab (600 mg fixed dose IV).
  * Ibrutinib self-administered orally QD, continuously starting concurrently with cirmtuzumab in Week 0 at a dose of either 420 mg/day (for patients with CLL/SLL) or at a dose of 560 mg/day (for patients with MCL or MZL).
- CLL Phase 2, Part 3: 600 mg; CLL Phase 2, Part 3: Ibrutinib Alone: Part 3 comprises a Phase 2 open-label, randomized, controlled, 2-arm, parallel-group evaluation of the clinical activity and safety of cirmtuzumab + ibrutinib versus ibrutinib alone. Patients with CLL/SLL will be randomized 2:1 to one of the following 2 regimens in blocks of 6 patients using a pre-generated randomization list:
  * Arm A: cirmtuzumab + ibrutinib
  * Arm B: ibrutinib alone
Period: Overall Study
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone
Started | 3 | 3 | 3 | 3 | 21 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 18 | 10
Efficacy Population CLL (Parts 1 & 2) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 0 | 0
Efficacy Population (Part 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 7
Efficacy Population MCL (Parts 1 & 2) | 3 | 3 | 3 | 3 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 21 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 18 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease Progression | 1 | 2 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Initiation of Alternative Treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 0
Not completed — Terminated by Sponsor | 2 | 1 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 3 | 13 | 2 | 1
Not completed — Completed 2 years of Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 8 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — COVID Related noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Drug or Study Noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- CLL Phase 1b, Part 2: 600 mg: Part 1:
  * Cirmtuzumab given by IV infusion every 2 weeks for 5 administrations (Weeks 0, 2, 4, 6, 8) and then every 4 weeks thereafter (Weeks 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52) at a dose of either 2, 4, 8, or 16 mg/kg. After establishment of safety at these dose levels, fixed doses of 300 and 600 mg IV per dose will be examined in patients with CLL/SLL.
  * Ibrutinib self-administered orally, QD, continuously starting in Week 4 at a dose of either 420 mg/day (for patients with CLL/SLL) or at a dose of 560 mg/day (for patients with MCL).
  Part 2:
  * Cirmtuzumab given by IV infusion every 2 weeks for 3 administrations (Weeks 0, 2, 4) and then every 4 weeks thereafter (Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52) using the RDR of cirmtuzumab (600 mg fixed dose IV).
  * Ibrutinib self-administered orally QD, continuously starting concurrently with cirmtuzumab in Week 0 at a dose of either 420 mg/day (for patients with CLL/SLL) or at a dose of 560 mg/day (for patients with MCL or MZL).
- Total: Total of all reporting groups
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600 mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 21 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 18 | 10 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (2.1) | 63.7 (6.0) | 59.0 (8.7) | 56.7 (11.6) | 66.6 (9.3) | 62.3 (7.6) | 74.0 (13.1) | 71.3 (8.1) | 68.7 (9.0) | 74.0 (2.7) | 71.3 (4.9) | 64.3 (9.5) | 66.2 (9.2) | 64.7 (6.7) | 66.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 4 | 0 | 3 | 0 | 0 | 1 | 0 | 4 | 8 | 7 | 29
  Male | 2 | 3 | 2 | 3 | 17 | 3 | 0 | 3 | 3 | 2 | 3 | 12 | 10 | 3 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4
  White | 2 | 3 | 1 | 2 | 18 | 2 | 2 | 3 | 3 | 3 | 1 | 15 | 15 | 8 | 78
  More than one race | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 21 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 18 | 10 | 95

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Defined as achievement of complete response (CR), complete response with incomplete blood count recovery (CRi), partial response (PR), or partial response with lymphocytosis (PR-L) for those with CLL/SLL, per standardized criteria [Hallek 2008], as recently updated [Hallek 2018; Cheson 2012]; and the achievement of a CR or PR for those with MCL or MZL, per based on standardized criteria [Cheson 2007] as recently updated [Cheson 2014].
Time Frame: up to 5 years
Population: The efficacy population consists of enrolled subjects who have received at least one dose of either cirmtuzumab or ibrutinib and at least one tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 16 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 7
Participants | 3 | 3 | 3 | 2 | 14 | 3 | 3 | 2 | 3 | 3 | 2 | 15 | 15 | 7

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression or death from any cause. PFS was analyzed using Kaplan-Meier Survival Methods.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 16 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 7
months | NA [35.9 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [16.5 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | 4.3 [0.03 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | 36.3 [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [15.7 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [41.6 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [25.9 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. | NA [11.0 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI.

3. Secondary Outcome: Overall Survival
Description: Defined as the interval from the start of study therapy to death from any cause. Overall Survival was analyzed using Kaplan-Meier Survival methods.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 16 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 7
months | NA [NA to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [18.8 to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | 22.5 [11.5 to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [14.0 to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [36.3 to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [15.7 to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [41.6 to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [19.7 to NA] — NA for median indicates that there were not enough OS events (i.e., death) to estimate the median time to OS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results.

4. Secondary Outcome: Duration of Response
Description: Defined as the amount of time (months) for achieving of complete response (CR), complete response with incomplete blood count recovery (CRi), partial response (PR), or partial response with lymphocytosis (PR-L) for those with CLL/SLL; and the amount of time (months) for achieving of a CR or PR for those with MCL.
Time Frame: Up to 5 years
Population: The subset of the efficacy population achieving Objective Response (ORR). The efficacy population consists of enrolled subjects who have received at least one dose of either cirmtuzumab or ibrutinib and at least one tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 14 | 3 | 3 | 2 | 3 | 3 | 2 | 15 | 15 | 7
months | NA [34.1 to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [13.8 to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | 11.9 [1.5 to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | 33.5 [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | 38.8 [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | 40.3 [19.6 to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [22.2 to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [8.3 to NA] — NA for median indicates that there were not enough Duration of Response events (i.e., progressive disease or death) to estimate the median time to Duration of Response (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results.

5. Secondary Outcome: Progression-free Survival (PFS) for Patients With TP53 Mutation Status
Description: Defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression or death from any cause, in patients with TP53 mutation status
Time Frame: Up to 5 years
Population: A subset of the efficacy population with a positive Del(17p) mutation. The efficacy population consists of enrolled subjects who have received at least one dose of either cirmtuzumab or ibrutinib and at least one tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 3 | 1
months |  | 16.5 [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | 17.3 [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. |  | NA [2.8 to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. |  |  |  |  | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. |  | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results. | NA [NA to NA] — NA for median indicates that there were not enough PFS events (i.e., progressive disease or death) to estimate the median time to PFS (i.e. 50% Survival). NA for the 95% CI limits indicates that there were not enough events above/below the 50% survival proportion to estimate the limit of the CI. Kaplan-Meier Survival methods were used for reporting analysis results.

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | MCL Phase 1b, Part 1: 2mg/kg | MCL Phase 1b, Part 1: 4mg/kg | MCL Phase 1b, Part 1: 8mg/kg | MCL Phase 1b, Part 1: 16 mg/kg | MCL Phase 1b, Part 2: 600 mg | CLL Phase 1b, Part 1: 2 mg/kg | CLL Phase 1b, Part 1: 4 mg/kg | CLL Phase 1b, Part 1: 8 mg/kg | CLL Phase 1b, Part 1: 16 mg/kg | CLL Phase 1b, Part 1: 300 mg | CLL Phase 1b, Part 1: 600 mg | CLL Phase 1b, Part 2: 600 mg | CLL Phase 2, Part 3: 600 mg | CLL Phase 2, Part 3: Ibrutinib Alone
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 3/3 | 1/3 | 7/21 | 1/3 | 0/3 | 1/3 | 0/3 | 1/3 | 0/3 | 1/16 | 3/18 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 0/3 | 2/3 | 13/21 | 3/3 | 1/3 | 2/3 | 1/3 | 2/3 | 2/3 | 5/16 | 9/18 | 5/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 21/21 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 15/16 | 18/18 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCL Phase 1b, Part 1: 2mg/kg (N=3) | MCL Phase 1b, Part 1: 4mg/kg (N=3) | MCL Phase 1b, Part 1: 8mg/kg (N=3) | MCL Phase 1b, Part 1: 16 mg/kg (N=3) | MCL Phase 1b, Part 2: 600 mg (N=21) | CLL Phase 1b, Part 1: 2 mg/kg (N=3) | CLL Phase 1b, Part 1: 4 mg/kg (N=3) | CLL Phase 1b, Part 1: 8 mg/kg (N=3) | CLL Phase 1b, Part 1: 16 mg/kg (N=3) | CLL Phase 1b, Part 1: 300 mg (N=3) | CLL Phase 1b, Part 1: 600 mg (N=3) | CLL Phase 1b, Part 2: 600 mg (N=16) | CLL Phase 2, Part 3: 600 mg (N=18) | CLL Phase 2, Part 3: Ibrutinib Alone (N=10)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erosive Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypnonatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Respiratory Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular Disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial Haemorrhage (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atheroembolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eschericha Urinary Tract Infection (Infections and infestations) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCL Phase 1b, Part 1: 2mg/kg (N=3) | MCL Phase 1b, Part 1: 4mg/kg (N=3) | MCL Phase 1b, Part 1: 8mg/kg (N=3) | MCL Phase 1b, Part 1: 16 mg/kg (N=3) | MCL Phase 1b, Part 2: 600 mg (N=21) | CLL Phase 1b, Part 1: 2 mg/kg (N=3) | CLL Phase 1b, Part 1: 4 mg/kg (N=3) | CLL Phase 1b, Part 1: 8 mg/kg (N=3) | CLL Phase 1b, Part 1: 16 mg/kg (N=3) | CLL Phase 1b, Part 1: 300 mg (N=3) | CLL Phase 1b, Part 1: 600 mg (N=3) | CLL Phase 1b, Part 2: 600 mg (N=16) | CLL Phase 2, Part 3: 600 mg (N=18) | CLL Phase 2, Part 3: Ibrutinib Alone (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 6 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 3 (6) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 5 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (7) | 1 (1) | 3 (5) | 3 (6) | 9 (14) | 1 (5) | 2 (3) | 1 (2) | 1 (3) | 1 (1) | 1 (2) | 8 (16) | 5 (7) | 5 (8)
Fatigue (General disorders) | 3 (7) | 3 (4) | 2 (2) | 1 (1) | 7 (7) | 2 (4) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (2) | 7 (9) | 6 (12) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03088878/Prot_SAP_002.pdf